CLINICAL TRIAL: NCT07401602
Title: A Retrospective Evaluation of Systemic Analgesia, Rhomboid Intercostal Block, and Combined Rhomboid Intercostal Block With Deep Parasternal Intercostal Plane Block After Mastectomy
Brief Title: Analgesic Strategies After Mastectomy: RIB vs RIB + DPIPB
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, associate professor, Istinye University
Other Study IDs: zeki mastektomi
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Systemic Analgesia Group
  Interventions: Other: Analgesic Strategy
- Rhomboid Intercostal Block (RIB) Group
  Interventions: Other: Analgesic Strategy
- RIB + Deep Parasternal Intercostal Plane Block (DPIPB) Group
  Interventions: Other: Analgesic Strategy

INTERVENTIONS:
Other: Analgesic Strategy — Systemic Analgesia:
  Postoperative pain was managed using standard systemic analgesic medications as part of routine clinical care.
  Rhomboid Intercostal Block (RIB):
  Postoperative analgesia was provided using an ultrasound-guided rhomboid intercostal block performed as part of routine clinical practice.
  RIB + Deep Parasternal Intercostal Plane Block (DPIPB):
  Postoperative analgesia was provided using a combination of ultrasound-guided rhomboid intercostal block and deep parasternal intercostal plane block as part of routine clinical care.

SUMMARY:
This retrospective observational study evaluates postoperative pain outcomes in patients undergoing elective mastectomy who received systemic analgesia, rhomboid intercostal block (RIB), or combined rhomboid intercostal block with deep parasternal intercostal plane block (RIB + DPIPB). Medical records from October 2024 to October 2025 will be reviewed. Primary outcomes include pain scores within the first 24 hours, with secondary outcomes including opioid consumption, additional analgesic requirements, patient satisfaction, and early postoperative complications. All data will be analyzed retrospectively and anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-70 years
* Elective mastectomy performed between October 2024 and October 2025
* ASA physical status I-III
* Complete postoperative pain and analgesia records for the first 24 hours
* Clearly documented analgesic technique (systemic analgesia, RIB, or RIB + DPIPB)

Exclusion Criteria:

* Incomplete or missing medical records
* Emergency mastectomy or emergency surgery
* Reoperation within the first 24 hours postoperatively
* Major intraoperative complications preventing standard analgesia
* Neurological or psychiatric conditions interfering with pain assessment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult female patients aged 18-70 years who underwent elective mastectomy at a single tertiary care center between October 2024 and October 2025 and had complete postoperative pain and analgesia records available for retrospective analysis.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score (VAS) | Within the first 24 hours after surgery (postoperative 1, 6, 12, and 24 hours).
  Postoperative pain intensity assessed using the Visual Analog Scale (VAS) based on routinely recorded clinical data.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Result] Ertas G, Cakmak HS, Ocak S, Yilmaz M, Ozdemir DB, Tulgar S. Is the combination of interfascial plane blocks sufficient for awake breast cancer surgery? An observational, prospective, proof-of-concept study. BMC Anesthesiol. 2024 Sep 20;24(1):337. doi: 10.1186/s12871-024-02725-0. PMID 39304815
- [Result] Gu B, Huang ZX, Zhou HD, Lian YH, He S, Ge M, Jiang HF. A Randomized Controlled Trial of Adding Deep Parasternal Intercostal Plane Block to Interpectoral-Pectoserratus Plane Block in Breast Cancer Surgery. Anesth Analg. 2025 May 1;140(5):1188-1194. doi: 10.1213/ANE.0000000000007218. PMID 39453840